CLINICAL TRIAL: NCT07231965
Title: Effects Of Cannabis Products On Blood Pressure Control
Brief Title: Synthetic THC And Blood Pressure
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25-008291
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dronabinol Group (Active Comparator): Patients taking Dronabinol first and Placebo second
  Interventions: Drug: Dronabinol; Drug: Placebo
- Placebo Group (Active Comparator): Patients taking Placebo first and Dronabinol second
  Interventions: Drug: Dronabinol; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Patients will take one 10 mg dose of Dronabinol.
Drug: Placebo — Patients will take one 10mg dose of a Placebo Pill.

SUMMARY:
To investigate the effects of Dronabinol use on blood pressure and neurovascular physiology

ELIGIBILITY:
Inclusion Criteria

* Recreational occasional Cannabis use (Consuming THC less than 2 times a week)
* 21 - 40 years of age
* Biological male or female

Exclusion Criteria

* BMI > 35 kg/m2
* Diagnosed psychiatric disorders
* Hypotension
* History of seizures
* History of substance abuse or recreational drug use or positive urine drug screen
* History of uncontrolled disease including:

  * Cardiovascular
  * Pulmonary
  * Gastrointestinal
  * Pancreatic
  * Hepatic
  * Renal
  * Hematological
  * Endocrine (including Type I Diabetes)
  * Neurological
  * Urological
  * Sleep disorders
* Pregnant or breastfeeding
* Use of certain antimicrobial, chemotherapeutic, anticoagulant, hypoglycemic, anti-inflammatory, psychotropic, and antihistamine drugs
* Prescribed CYP2C9 and/or CYP3A4 inhibitors
* History of shift work or rotating shifts within 1 month

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, 30 days
  Blood pressure is the force exerted by circulating blood on the walls of the arteries as it is pumped through the body. Blood pressure will be measured as a ratio of systolic/diastolic (mmHg).
Heart Rate | Baseline, 30 days
  Heart Rate is the number of contractions (beats) that the heart makes per minute. This will be measured in bpm (beats per minute)

SECONDARY OUTCOMES:
Baroreflex Sensitivity | Baseline, 30 days
  Baroreflex sensitivity will be assessed using beat-by-beat blood pressure, heart rate, and Sympathetic nerve activity collected continuously for at least 5min. This will be measured in ms/mmHg.
Sympathetic control | Baseline, 30 days
  Sympathetic control will be measured by microneurography of peroneal or fibular nerve, reported as bursts of sympathetic activity per minute or normalized to 100 heart beats
Flow Mediated Dilation | Baseline, 30 days
  Flow Mediated Dilation will be measured by ultrasonography of brachial artery, reported as an absolute change in arterial diameter from resting baseline
Aortic Wave Reflection | Baseline, 30 days
  Aortic Wave Reflection will be measured via arterial tonometry, reported as aortic augmentation index

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No